CLINICAL TRIAL: NCT05884827
Title: Peroneal Nerve Dysfunction in Proximal Fibular Epiphyseal Harvesting Cases
Brief Title: Peroneal Nerve Dysfunction in Epiphyseal Transfer
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Moustafa Elsese, Principal investigator, Assiut University
Other Study IDs: EMG in Epiphyseal transfer
Record Dates: First submitted 2023-04-23; First posted 2023-06-01 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Epiphyseal Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EMG — Measure the electrical activity of the muscle and nerve

SUMMARY:
Assessment of peroneal nerve dysfunction after proximal fibular epiphyseal resection and evaluation of clinical outcome and EMG changes.

DETAILED DESCRIPTION:
In children the preserved epiphysis of the proximal fibula ensure the exceptional ability to recover both joint function and longitudinal limb growth at the same time. Traumatic bone defect, congenital malformations, malignant bone lesions and infection are all current indications for VFET. The shape and size of the proximal fibular epiphysis aid in the gradual remodeling of the articular surface, allowing for better reconstruction and eventual rehabilitation over time.

Harvesting the proximal epiphysis of the fibula, along with its intact blood supply, is technically demanding, and the success of VFET is a primarily dependent on restoring adequate vascularity to the growth plate and diaphysis.

Anterior tibial artery is the primary and most consistent contributor to the proximal fibular epiphysis and proximal two thirds of diaphysis, it has intimate connection to the motor (deep) branch of peroneal nerve. The success of anterior tibial artery based VFET based on preserving the anterior tibial Vascular bundle, so it may be necessary to sacrifice some branches of peroneal nerve to tibialis anterior muscle. This is a significant flaw in the approach that could result in permanent peroneal nerve palsy.

ELIGIBILITY:
Inclusion Criteria:

* all patients candidate for epiphyseal transfer are included ( patients with traumatic bone defect, congenital malformations, malignant bone lesions and infection )

Exclusion Criteria:

* patients in which there's no injury of nerve supply of tibialis anterior has occurred intraoperative

Ages: 18 Months to 14 Years | Sex: All
Age Groups: Child
Study Population: Children with destroyed epiphysis whatever the cause of destruction and with preserved proximal fibular epiphysis
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of Tibialis anterior dysfunction after proximal fibular epiphyseal harvesting | Six months
  Electromyography changes at 3 weeks , 6 weeks , 3 months and 6 months to assess the affection of tibialis anterior muscle & peroneal nerve

CONTACTS AND LOCATIONS:
Locations (1):
- Omar, Asyut, Egypt

REFERENCES:
- [Background] Zelenski N, Brigman BE, Levin LS, Erdmann D, Eward WC. The vascularized fibular graft in the pediatric upper extremity: a durable, biological solution to large oncologic defects. Sarcoma. 2013;2013:321201. doi: 10.1155/2013/321201. Epub 2013 Oct 7. PMID 24222724
- [Background] Shammas RL, Avashia YJ, Farjat AE, Catanzano AA, Levin LS, Eward WC, Brigman BE, Erdmann D. Vascularized Fibula-Based Physis Transfer: A Follow-Up Study of Longitudinal Bone Growth and Complications. Plast Reconstr Surg Glob Open. 2017 May 25;5(5):e1352. doi: 10.1097/GOX.0000000000001352. eCollection 2017 May. PMID 28607872
- [Background] Ghert M, Colterjohn N, Manfrini M. The use of free vascularized fibular grafts in skeletal reconstruction for bone tumors in children. J Am Acad Orthop Surg. 2007 Oct;15(10):577-87. doi: 10.5435/00124635-200710000-00001. PMID 17916780
- [Background] Innocenti M, Delcroix L, Romano GF. Epiphyseal transplant: harvesting technique of the proximal fibula based on the anterior tibial artery. Microsurgery. 2005;25(4):284-92. doi: 10.1002/micr.20130. PMID 15934045
- [Background] Sales de Gauzy J, Accadbled F, Gomez Brouchet A, Abid A. Case report: histologic study of a human epiphyseal transplant at 3 years after implantation. Clin Orthop Relat Res. 2009 Jul;467(7):1915-20. doi: 10.1007/s11999-009-0723-z. Epub 2009 Feb 11. PMID 19212796
- [Background] Grimer RJ. Surgical options for children with osteosarcoma. Lancet Oncol. 2005 Feb;6(2):85-92. doi: 10.1016/S1470-2045(05)01734-1. PMID 15683817